CLINICAL TRIAL: NCT00955084
Title: A Maintenance Study Evaluating the Long Term Safety of XL999 Administered Intravenously to Subjects With Advanced Malignancies Previously Enrolled in Other XL999 Studies
Brief Title: Maintenance Study on the Long Term Safety of XL999
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W Finn, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-900
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: XL999 — XL999 for injection will be supplied as a brown, sterile injectable solution at a concentration of 5 mg/mL

SUMMARY:
The primary objective of this study is to allow rollover of the two remaining subjects from the other XL999 studies to continue to receive XL999.

The secondary objectives of this study are as follows:

* To evaluate tumor response after long term repeat administration of XL999 in two subjects rolled over from other XL999 studies.
* To characterize the long term safety and tolerability of XL999 after repeat administration in two subjects rolled over from other XL999 studies.
* To characterize the long term effects of XL999 on cardiac function after repeat administration in two subjects rolled over from other XL999 studies.

ELIGIBILITY:
Inclusion Criteria:

* The subject is currently enrolled in Protocols XL999-001 or XL999-204
* The subject has received XL999 for at least one year prior to enrollment
* Per the respective parent XL999 protocol, the subject is eligible to continue to receive XL999 in the absence of progressive disease (PD) or unacceptable drug-related toxicity

Exclusion Criteria:

* Progressive disease
* Any development(s) that would meet the exclusion criteria from the subject's respective XL999 protocol (XL999-001 or XL999-204)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to allow rollover of the two remaining subjects from the other XL999 studies to continue to receive XL999. | Progressive disease or end of study

SECONDARY OUTCOMES:
Evaluate tumor response after long term repeat administration of XL999 Characterize long term safety and tolerability of XL999 after repeat administration Characterize long term effects of XL999 on cardiac function after repeat administration | Progressive disease or end of study

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Finn, PhD, Study Director — Symphony Evolution, Inc.
Locations (2):
- United States (2):
  - Hematology Oncology Associates of Rockland Union State Bank Cancer Center, Nyack, New York
  - University of Texas Cancer Center, San Antonio, Texas